CLINICAL TRIAL: NCT05821296
Title: Evaluation of the Efficacy and Tolerance of Crystal Peel (a Salicylic Acid Based Peel) in the Treatment of Acne
Brief Title: Evaluation of Efficacy and Tolerance of Crystal Peel in the Treatment of Adults Presenting Facial Mild Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dermosciences France (Industry)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22E2387
Record Dates: First submitted 2023-02-03; First posted 2023-04-20 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Acne Vulgaris
Keywords: acne; facial; crystal peel; salicylic acid; chemical peel
MeSH Terms: conditions — Acne Vulgaris; Facies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Crystal Peel (Other): 2.5 ml of Crystal peel applied up to 3 coats and performed 3 times in the study (i.e: at Day 15, Day 36 and Day 57.
  Interventions: Device: Crystal Peel

INTERVENTIONS:
Device: Crystal Peel — 3 applications performed by a dermatologist.

SUMMARY:
The goal of this interventional, confirmatory and post market study is to evaluate the efficacy and clinical performance of Crystal Peel in adults suffering mild facial acne vulgaris. The principal and secondary aims are:

* Principal aim: to evaluate the efficacy and clinical performance of Crystal Peel, a salicylic-based peel, for the treatment of acne by lesions counting (front, 2 cheeks, the chin above the jaw line (excluding the nose)) using both visual observation and palpation.
* Secondary aims: pores and texture analysis, visual effect (Standardized anonymized photographs, investigator global assessment, patient global assessment, local and overall tolerance of the Crystal Peel, subject's self-evaluation and potential adverse events collection.

The primary endpoint of the study will be an objective counting of the acne lesions performed on every visit.

DETAILED DESCRIPTION:
Total lesions will be defined as the sum of inflammatory lesions (papules and pustules), non-inflammatory lesions (whiteheads and blackheads) and other acne lesions (nodules).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects
2. Gender: female and/or male.
3. Age: 18 - 45
4. Phototype I to IV according Fitzpatrick scale.
5. Healthy subject with normal physical examination results and a medical history compatible with the requirements of the study.
6. A healthy male or female subject with a medical diagnosis of mild to moderate facial acne vulgaris defined by at least 6 (six) inflammatory lesions, 12 (twelve) non-inflammatory lesions and no more than 2 (two) nodules (the nose is excluded for lesion count purposes).
7. Subject declares to avoid exposure to UV radiation (tanning booths, phototherapy and sun) on the face for at least three months prior to the selection visit and agrees to avoid it throughout the study.
8. Subject agrees not to apply any cosmetic, medical or aesthetic treatments outside the study protocol on the face for the duration of the study.
9. For female subjects:

Female subject not in childbearing status (tubal ligation, hysterectomy, bilateral oophorectomy), or Female subjects of childbearing potential who, in the opinion of the investigator, are using a reliable method of contraception (pill or contraceptive patch, IUD, implant or vaginal ring,condoms) for at least one month prior to the screening visit. Subject willing to continue using contraception during the study and one month after the end of the study.

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
3. Subject in a social or sanitary establishment.
4. Subject participating to another clinical research or being in an exclusion period for a previous study.
5. Intensive exposure to sunlight or UV-rays within the previous 3 months and foreseen during the study.
6. Subject with any skin or systemic disease (acute and/or chronic), in the previous year, likely to interfere with the measured parameters or to put the subject to an undue risk.
7. Subject having history of allergy or hypersensitivity to one of the components of the tested device.
8. Subject receiving any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject to undue risk.
9. Subjects on topical or oral treatments (such as Benzoyl Peroxide, Retinoic Acid, isotretinoin) that did not stop the treatment 30 days before their first peel (risk of over-peeling).
10. Subjects with known salicylism or related medical indications.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beata IMKO-WALCZUK, Dr, Principal Investigator — Eurofins Dermscan Poland
Locations (1):
- Eurofins Dermscan Poland, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on dermatologist referral in a single-site between January 2023 and March 2023.
  The first patient was enrolled on January 23, 2023 and the last patient was enrolled on March 3, 2023.
Pre-assignment Details: Of 42 enrolled patients, 33 met study eligibility criteria and were included to Crystal Peel treatment and 9 did not met inclusion criteria number 6 (i.e: low number of acne lesions).
Groups:
- Crystal Peel: Patients received 2.5 ml of Crystal peel topically applied up to 3 coats and performed 3 times in the study (i.e: at Day 15, Day 36 and Day 57).
  Crystal Peel: 3 applications performed by a dermatologist.
Period: Overall Study
Arm/Group | Crystal Peel
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 33
Fitzpatrick skin phototype [Number; unit: participants] — Fitzpatrick skin phototypes (from I to IV) used to characterize studied population. For guidance on Fitzpatrick skin phototypes, (Rünger 2019).
  I: always burns, never tans. Pale white color of unexposed skin. II: always burns, then tans. White color of unexposed skin. III: sometimes burns, can tan without prior burn. White color of unexposed skin.
  IV: usually does not burn, tans easily and deeply. White to light brown color of unexposed skin.
  participants
    Skin phototype I | 0
    Skin phototype II | 26
    Skin phototype III | 7
    Skin phototype IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Change From Baseline of Count Lesions on Each Visit to Evaluate the Efficacy and Clinical Performance of Crystal Peel for the Treatment of Acne.
Description: Lesion counting using both visual observation and palpation. Total lesions (front, 2 cheeks, the chin above the jaw line (excluding the nose)) will be defined as the sum of inflammatory lesions (papules, pustules), non-inflammatory lesions (whiteheads and blackheads) and other acne lesions (nodules).
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: Per protocol (PP) population (any patient having used at least once the investigational device and without any major deviation to the clinical investigation plan.
Measure: Count of Units; unit: Lesions count at each protocol visit
Units Other Than Participants: Lesions count at each protocol visit
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
Number analyzed (Lesions count at each protocol visit) | 943
Lesions count at each protocol visit
  Lesions count at Day 0 | 943
  Lesions count at Day 15 | 647
  Lesions count at Day 36 | 457
  Lesions count at Day 57 | 407
  Lesions count at Day 78 | 463
Statistical Analysis 1: Comparison: Crystal Peel; Test type: Other — Change of sum of total lesions at the end of the study from baseline/Day 0 to evaluate the efficacy and clinical performance of Crystal Peel for the treatment of acne; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.58, 95% CI 2-sided [-17.31 to -11.84], Standard Error of Mean 1.38

2. Secondary Outcome: Acne Investigator Global Assessment (IGA) Score
Description: Investigator's global assessment of acne condition improvement at Day 78 (last protocol visit). The score range is -1 to 3, with higher scores denoting better outcomes, better acne condition improvement from baseline. Score ranges details: -1 (worse), 0 (no improvement), 1 (good improvement), 2 (very good improvement) on Day 78 (last protocol visit).
Time Frame: At Visit 5/Day 78.
Population: Per protocol (PP) population (any patient having used at least once the investigational device and without any major deviation to the clinical investigational plan).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Crystal Peel: 2.5 ml of Crystal peel applied up to 3 coats and performed 3 times in the study (i.e: at Day 15, Day 36 and Day 57).
  Crystal Peel: 3 applications performed by a dermatologist.
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
score on a scale | 1.85 (0.87)
Statistical Analysis 1: Comparison: Crystal Peel; Test type: Other; Mean Difference (Final Values) = 1.85, 95% CI 2-sided [1.54 to 2.16], Standard Deviation 0.87

3. Secondary Outcome: Acne Patient Global Assessment (PGA) Scale
Description: Patient's global assessment of acne condition improvement at Day 78 (last protocol visit). The score range is -1 to 3, with higher scores denoting better outcomes, better acne condition improvement from baseline. Score ranges details: -1 (worse), 0 (no improvement), 1 (good improvement), 2 (very good improvement) on Day 78 (last protocol visit).
Time Frame: At Visit 5/Day 78.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
score on a scale | 1.82 (1.07)
Statistical Analysis 1: Comparison: Crystal Peel; Test type: Other; Mean Difference (Final Values) = 1.82, 95% CI 2-sided [1.44 to 2.20], Standard Deviation 1.07

4. Secondary Outcome: Local and Overall Tolerance of the Crystal Peel.
Description: At the end of the study, the local tolerance on the skin of the product has been assessed during the clinical examination by the investigator by the "Local tolerance scale" (from 0 to 3, where higher scores mean better outcome) according to the following scores: 0= bad tolerance; 1= moderate tolerance; 2= good tolerance and 3= very good tolerance.
Time Frame: At Visit 5/Day 78).
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
Participants
  Very good tolerance | 10
  Good tolerance | 21
  Moderate tolerance | 1
  Bad tolerance | 1
Statistical Analysis 1: Comparison: Crystal Peel; Test type: Other; Mean value in local tolerance score = 2.21, 95% CI 2-sided [1.98 to 2.44], Standard Deviation 0.65

5. Secondary Outcome: Subject's Satisfaction Questionnaire
Description: Count and percentage of subjects who answered satisfactorily to the 17-item questionnaire that measured patients' satisfaction after use of Crystal Peel in treating acne at Day 78 (final protocol visit).
Time Frame: At Visit 5/Day 78.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
Participants
  The treatment you tried prevented your acne from getting worse | 26
  The treatment you have experienced has reduced the surface area of your acne | 31
  Blemishes are visibly reduced | 29
  Pores are tightened and less visible | 31
  Skin texture is improved | 28
  The skin is matified | 30
  The skin is clearer | 30
  Satisfactory effectiveness of this treatment | 28
  This treatment is of high performance | 26
  I am delighted with the results obtained to date | 26
  The treatment met my needs | 29
  The treatment is not restrictive | 28
  Compared to other treatments, this one is more effective | 25
  Thanks to this treatment, I feel better in my skin | 28
  I would like to continue this treatment | 33
  I will be interested in renewing this treatment with a practitioner | 33
  I will advise someone else to use this treatment | 33
Statistical Analysis 1: Comparison: Crystal Peel; Test type: Other — Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; % of patients with positive answers = 79, 95% CI 2-sided [61 to 89]
Statistical Analysis 2: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 94, 95% CI 2-sided [80 to 98]
Statistical Analysis 3: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 88, 95% CI 2-sided [73 to 95]
Statistical Analysis 4: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 85, 95% CI 2-sided [68 to 93]
Statistical Analysis 5: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 91, 95% CI 2-sided [77 to 97]
Statistical Analysis 6: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 85, 95% CI 2-sided [69 to 93]
Statistical Analysis 7: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 78, 95% CI 2-sided [61 to 89]
Statistical Analysis 8: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 79, 95% CI 2-sided [62 to 89]
Statistical Analysis 9: Comparison: Crystal Peel; Descriptive analysis of subjects' satisfaction questionnaire assessing the Crystal Peel in the treatment of acne; Test type: Other; % of patients with positive answers = 76, 95% CI 2-sided [59 to 87]

6. Secondary Outcome: Number of Adverse Events
Description: Collection of adverse events by the investigator. Please refer to Adverse Events tables for more details.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: Safety population: any subject having used the investigational device. 33 patients have been analyzed.
Measure: Number; unit: adverse events
Units Other Than Participants: adverse events
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
Number analyzed (adverse events) | 217
adverse events
  Adverse events not related to studied product : mild | 92
  Adverse events not related to studied product : moderate | 22
  Adverse events not related to studied product : severe | 0
  Adverse events related to studied product : mild | 103
  Adverse events related to studied product : moderate | 0
  Adverse events related to studied product : severe | 0

7. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Number of Detected Pores on Each Visit to Evaluate the Improvement of Pores Assessed by Colorface Device.
Description: Front face image with parallel polarization will be analyzed. A region of interest is defined on the cheek near the nose of each subject at baseline, it has the same size for all subjects and is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous number is defined as the number of distinct elements in the segmentation. A decrease of the conspicuous number of pores results in a decrease of the number of pores that are detected by the algorithm. There is an improvement of pores if and only if one of the following parameters is decreasing and the other ones are stable (no statistically significance) or decreasing: conspicuous number, conspicuous area, average area, conspicuous density, conspicuous depth and conspicuous volume of detected pores.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of detected pores
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
number of detected pores
  Conspicuous number of detected pores at Day 0 | 355.03 (133.03)
  Conspicuous number of detected pores at Day 15 | 307.79 (133.99)
  Conspicuous number of detected pores at Day 36 | 324.18 (133.92)
  Conspicuous number of detected pores at Day 57 | 309.34 (110.80)
  Conspicuous number of detected pores at Day 78 | 321.91 (123.81)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous number of detected pores at day 15 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p < 0.0001, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Net) = -47.24, Standard Deviation 56.61
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous number of detected pores at Day 36 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.010, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -30.85, Standard Deviation 63.92
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous number of detected pores at Day 57 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p < 0.004, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -41.69, Standard Deviation 73.69
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous number of detected pores at day 78 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.013, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -29.13, Standard Deviation 61.45

8. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Area of Detected Pores on Each Visit to Evaluate the Improvement of Pores Assessed by Colorface Device.
Description: Front face image with parallel polarization will be analyzed. A region of interest is defined on the cheek near the nose of each subject at baseline, it has the same size for all subjects and is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous area is defined as the total number of pixels in the segmentation (total surface of detected pores). A decrease of the conspicuous area results in a decrease of the total surface occupied by detected pores. There is an improvement of pores if and only if one of the following parameters is decreasing and the other ones are stable (no statistically significance) or decreasing: conspicuous number, conspicuous area, average area, conspicuous density, conspicuous depth and conspicuous volume of detected pores.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: total number of pixels
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
total number of pixels
  conspicuous area of detected pores at Day 0 | 19088.48 (9179.66)
  conspicuous area of detected pores at Day 15 | 16256.09 (9179.12)
  conspicuous area of detected pores at Day 36 | 17333.61 (8895.27)
  conspicuous area of detected pores at Day 57 | 16109.97 (7666.83)
  conspicuous area of detected pores at Day 78 | 17130.97 (8546.22)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of detected pores at day 15 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p < 0.0001, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -2832.39, Standard Deviation 3217.15
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of detected pores at day 36 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.025, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -1754.88, Standard Deviation 4220.25
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of detected pores at day 57 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.004, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -2763.41, Standard Deviation 4965.84
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of detected pores at day 78 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.021, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -1742.41, Standard Deviation 3974.21

9. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Relative Area (Density) of Detected Pores on Each Visit to Evaluate the Improvement of Pores Assessed by Colorface Device.
Description: Front face image with parallel polarization will be analyzed. A region of interest is defined on the cheek near the nose of each subject at baseline, it has the same size for all subjects and is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm.The relative area is defined as the area of segmentation divided by total area of the region of interest. A decrease of conspicuous relative area results in a decrease of the detected pores conspicuous density. There is an improvement of pores if and only if one of the following parameters is decreasing and the other ones are stable (no statistically significance) or decreasing: conspicuous number, conspicuous area, average area, conspicuous density, conspicuous depth and conspicuous volume of detected pores.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
percentage
  Conspicuous relative area (density) of detected pores at Day 0 | 7.88 (3.23)
  Conspicuous relative area (density) of detected pores at Day 15 | 6.69 (3.32)
  Conspicuous relative area (density) of detected pores at Day 36 | 7.21 (3.40)
  Conspicuous relative area (density) of detected pores at Day 57 | 6.82 (3.01)
  Conspicuous relative area (density) of detected pores at Day 78 | 7.23 (3.37)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous relative area (density) of detected pores at Day 15 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p < 0.0001, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -1.20, Standard Deviation 1.30
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous relative area (density) of detected pores at Day 36 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.029, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.68, Standard Deviation 1.68
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous relative area (density) of detected pores at Day 57 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.006, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -1.07, Standard Deviation 2.01
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous relative area (density) of detected pores at Day 78 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.037, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Net) = -0.65, Standard Deviation 1.67

10. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Depth of Detected Pores on Each Visit to Evaluate the Improvement of Pores Assessed by Colorface Device.
Description: Front face image with parallel polarization will be analyzed. A region of interest is defined on the cheek near the nose of each subject at baseline, it has the same size for all subjects and is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous depth is defined as the difference of intensity between detected pores segmentation and surrounding segmentation. It is an average value over the whole region of interest. A decrease of conspicuous depth results in a decrease of detected pores visibility. There is an improvement of pores if and only if one of the following parameters is decreasing and the other ones are stable (no statistically significance) or decreasing: conspicuous number, conspicuous area, average area, conspicuous density, conspicuous depth and conspicuous volume of detected pores.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
arbitrary unit
  Conspicuous depth of detected pores at Day 0 | 7.12 (0.98)
  Conspicuous depth of detected pores at Day 15 | 6.73 (1.03)
  Conspicuous depth of detected pores at Day 36 | 6.98 (1.10)
  Conspicuous depth of detected pores at Day 57 | 6.85 (1.05)
  Conspicuous depth of detected poresat Day 78 | 7.01 (1.23)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of detected pores at Day 15 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.001, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.39, Standard Deviation 0.58
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of detected pores at Day 36 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.348, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.14, Standard Deviation 0.71
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of detected pores at Day 57 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.091, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.27, Standard Deviation 0.75
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of detected pores at Day 78 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.190, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.12, Standard Deviation 0.65

11. Secondary Outcome: Comparison of Change From Baseline of Average Area of Detected Pores on Each Visit to Evaluate the Improvement of Pores Assessed by Colorface Device.
Description: Front face image with parallel polarization will be analyzed. A region of interest is defined on the cheek near the nose of each subject at baseline, it has the same size for all subjects and is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The average area is defined as the area of segmentation divided by the number of distinct elements in the segmentation. It represents the average area of one detected pore. A decrease of the average area results in a decrease of the average size of detected pores or remaining detected pores if number decreases. There is an improvement of pores if and only if one of the following parameters is decreasing and the other ones are stable (no statistically significance) or decreasing: conspicuous number, conspicuous area, average area, conspicuous density, conspicuous depth and conspicuous volume of detected pores.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of pixels
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
number of pixels
  Average area of detected pores at Day 0 | 51.39 (9.44)
  Average area of detected pores at Day 15 | 49.70 (8.93)
  Average area of detected pores at Day 36 | 50.76 (9.34)
  Average area of detected pores at Day 57 | 49.75 (8.37)
  Average area of detected pores at Day 78 | 50.44 (8.87)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of average area of detected pores at Day 15 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.011, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -1.69, Standard Deviation 3.55
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of average area of detected pores at Day 36 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.281, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.64, Standard Deviation 3.28
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of average area of detected pores at Day 57 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.060, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -1.57, Standard Deviation 4.46
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of average area of detected pores at Day 78 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.209, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -0.87, Standard Deviation 3.80

12. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Volume of Detected Pores on Each Visit to Evaluate the Improvement of Pores Assessed by Colorface Device.
Description: Front face image with parallel polarization will be analyzed. A region of interest is defined on the cheek near the nose of each subject at baseline, it has the same size for all subjects and is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous volume is defined as the multiplication of conspicuous area and conspicuous depth. A decrease of conspicuous volume results in a decrease of detected pores visibility. There is an improvement of pores if and only if one of the following parameters is decreasing and the other ones are stable (no statistically significance) or decreasing: conspicuous number, conspicuous area, average area, conspicuous density, conspicuous depth and conspicuous volume of detected pores.
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Crystal Peel
Number analyzed (Participants) | 33
arbitrary unit
  Conspicuous volume of detected pores at Day 0 | 143085.53 (83078.48)
  Conspicuous volume of detected pores at Day 15 | 116589.71 (78431.52)
  Conspicuous volume of detected pores at Day 36 | 128638.51 (83941.10)
  Conspicuous volume of detected pores at Day 57 | 116400.38 (69989.53)
  Conspicuous volume of detected pores at Day 78 | 128428.39 (84587.06)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of detected pores at Day 15 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p < 0.0001, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -26495.83, Standard Deviation 33223.60
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of detected pores at Day 36 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.073, t-test, 2 sided; Mean Difference (Final Values) = -14447.02, Standard Deviation 44054.48
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of detected pores at Day 57 to evaluate the improvement of pores assessed by Colorface device; Test type: Other — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; p = 0.008, t-test, 2 sided; Mean Difference (Final Values) = -25315.34, Standard Deviation 49884.67
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of detected pores at Day 78 to evaluate the improvement of pores assessed by Colorface device; Test type: Other; p = 0.071, t-test, 2 sided — If the test provides a p-value less than 0.05, there is a significant variation over time for the analyzed parameter; Mean Difference (Final Values) = -13287.34, Standard Deviation 39615.92

13. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Area of Line Marks on Each Visit to Evaluate the Improvement of Line Marks Assessed by Colorface Device.
Description: Profiles images with parallel polarization will be analyzed by colorface device. A region of interest is delimited on the cheek of each subject at baseline and it is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous total area is defined as the number of pixels in segmentation of detected line marks. A decrease of conspicuous area results in a decrease of the total size of cheek line marks. There is an improvement of line marks if and only if one of the following parameters is decreasing and others ones are stable (no statistically significance) or decreasing: conspicuous area (unit=number of pixels), conspicuous length (unit=number of pixels), conspicuous depth (unit=arbitrary unit) and conspicuous volume of line marks (unit=arbitrary unit).
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: Intent-to-treat (ITT) population: any subject included in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: number of pixels
Arm/Group | Crystal Peel
Number analyzed (Participants) | 32
number of pixels
  Conspicuous area of line marks at Day 0 | 44845.94 (32444.07)
  Conspicuous area of line marks at Day 15 | 37327.69 (27992.85)
  Conspicuous area of line marks at Day 36 | 37615.13 (24073.14)
  Conspicuous area of line marks at Day 57 | 34126.74 (21031.09)
  Conspicuous area of line marks at Day 78 | 43277.71 (31379.00)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of line marks at Day 15 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney) — If the Wilcoxon test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -7518.25, Standard Deviation 13340.45
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of line marks at Day 36 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.041, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = -7230.81, Standard Deviation 17547.60
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of line marks at Day 57 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = -9086.26, Standard Deviation 18306.64
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous area of line marks at Day 78 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.931, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 13, analysis 1]; Mean Difference (Final Values) = 64.71, Standard Deviation 14542.17

14. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Depth of Line Marks on Each Visit to Evaluate the Improvement of Line Marks Assessed by Colorface Device.
Description: Profiles images with parallel polarization will be analyzed by Colorface device. A region of interest is delimited on the cheek of each subject at baseline and it is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The average conspicuous depth is defined as the difference of intensity between segmentation and surrounding segmentation. A decrease of conspicuous depth results in a decrease of cheek line marks visibility. There is an improvement of line marks if and only if one of the following parameters is decreasing and others ones are stable (no statistically significance) or decreasing: conspicuous area (unit=number of pixels), conspicuous length (unit=number of pixels), conspicuous depth (unit=arbitrary unit) and conspicuous volume of line marks (unit=arbitrary unit).
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: Intent-to-treat (ITT) population: any subject included in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Crystal Peel
Number analyzed (Participants) | 32
arbitrary unit
  Conspicuous depth of line marks at Day 0 | 7.57 (0.87)
  Conspicuous depth of line marks at Day 15 | 7.21 (0.75)
  Conspicuous depth of line marks at Day 36 | 7.26 (0.86)
  Conspicuous depth of line marks at Day 57 | 7.19 (0.78)
  Conspicuous depth of line marks at Day 78 | 7.57 (0.91)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of line marks at Day 15 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.005, t-test, 2 sided — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -0.36, Standard Deviation 0.66
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of line marks at Day 36 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.035, t-test, 2 sided — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -0.32, Standard Deviation 0.80
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of line marks at Day 57 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.036, t-test, 2 sided — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -0.34, Standard Deviation 0.86
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous depth of line marks at Day 78 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.784, t-test, 2 sided — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = 0.04, Standard Deviation 0.77

15. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Length of Line Marks on Each Visit to Evaluate the Improvement of Line Marks Assessed by Colorface Device.
Description: Profiles images with parallel polarization will be analyzed by colorface device. A region of interest is delimited on the cheek of each subject at baseline and it is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous length is defined as the total number of pixels in the morphological skeleton of segmentation. The morphological skeleton is defined as the central element of unit width of segmentation of detected line marks. A decrease of conspicuous length results in a decrease of the cumulated length of detected cheek line marks. There is an improvement of line marks if and only if one of the following parameters is decreasing and others ones are stable (no statistically significance) or decreasing: conspicuous area (unit=number of pixels), conspicuous length (unit=number of pixels), conspicuous depth (unit=arbitrary unit) and conspicuous volume of line marks (unit=arbitrary unit).
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: Intent-to-treat (ITT) population: any subject included in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: number of pixels
Arm/Group | Crystal Peel
Number analyzed (Participants) | 32
number of pixels
  Conspicuous length of line marks at Day 0 | 14139.88 (10628.03)
  Conspicuous length of line marks at Day 15 | 11890.16 (8944.85)
  Conspicuous length of line marks at Day 36 | 11824.88 (7823.46)
  Conspicuous length of line marks at Day 57 | 10849.32 (6827.80)
  Conspicuous length of line marks at Day 78 | 13980.52 (10631.19)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous length of line marks at Day 15 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney); If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -2249.72, Standard Deviation 4466.14
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous length of line marks at Day 36 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.074, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -2315.00, Standard Deviation 6197.86
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous length of line marks at Day 57 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -2700.55, Standard Deviation 5962.30
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous length of line marks at Day 78 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.779, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = 430.65, Standard Deviation 5021.20

16. Secondary Outcome: Comparison of Change From Baseline of Conspicuous Volume of Line Marks on Each Visit to Evaluate the Improvement of Line Marks Assessed by Colorface Device.
Description: Profiles images with parallel polarization will be analyzed by colorface device. A region of interest is delimited on the cheek of each subject at baseline and it is automatically repositioned at other timepoints for the same subject, thanks to a spatial registration algorithm. The conspicuous volume is defined as the multiplication of conspicuous area and conspicuous depth. A decrease of conspicuous volume results in a decrease of cheek line marks visibility. There is an improvement of line marks if and only if one of the following parameters is decreasing and others ones are stable (no statistically significance) or decreasing: conspicuous area (unit=number of pixels), conspicuous length (unit=number of pixels), conspicuous depth (unit=arbitrary unit) and conspicuous volume of line marks (unit=arbitrary unit).
Time Frame: At each protocol visit (i.e: Visit 1/Day 0, Visit 2/Day 15, Visit 3/Day 36, Visit 4/Day 57 and Visit 5/Day 78).
Population: Intent-to-treat (ITT) population: any subject included in the study with at least a post-basal value.
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Crystal Peel
Number analyzed (Participants) | 32
arbitrary unit
  Conspicuous volume of line marks at Day 0 | 359983.52 (301542.58)
  Conspicuous volume of line marks at Day 15 | 284182.77 (237265.18)
  Conspicuous volume of line marks at Day 36 | 286465.65 (206832.97)
  Conspicuous volume of line marks at Day 57 | 254170.91 (169281.12)
  Conspicuous volume of line marks at Day 78 | 345909.82 (284856.86)
Statistical Analysis 1: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of line marks at Day 15 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -75800.75, Standard Deviation 142643.92
Statistical Analysis 2: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of line marks at Day 36 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.054, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -73517.86, Standard Deviation 197224.85
Statistical Analysis 3: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of line marks at Day 57 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.008, Wilcoxon (Mann-Whitney) — If the test provides a p-value less than 0.05, the variation is significant over time for the studied parameter; Mean Difference (Final Values) = -90424.89, Standard Deviation 198264.20
Statistical Analysis 4: Comparison: Crystal Peel; Comparison of change from baseline of conspicuous volume of line marks at Day 78 to evaluate the improvement of line marks assessed by Colorface device; Test type: Other; p = 0.779, t-test, 2 sided; Mean Difference (Final Values) = 1314.03

ADVERSE EVENTS:
Time Frame: 78 days.
Description: Adverse events collection came from patient's diary and regular investigator assessment.
Arm/Group | Crystal Peel
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 33/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crystal Peel (N=33)
Burning sensation (Skin and subcutaneous tissue disorders) | 32 (51)
Desquamation (Skin and subcutaneous tissue disorders) | 17 (17)
Dryness (Skin and subcutaneous tissue disorders) | 13 (18)
Erythema (Skin and subcutaneous tissue disorders) | 33 (52)
Itching (Skin and subcutaneous tissue disorders) | 5 (6)
Sensation of coolness after peel application (Skin and subcutaneous tissue disorders) | 1 (1)
Skin tightness (Skin and subcutaneous tissue disorders) | 12 (20)
Stinging (Skin and subcutaneous tissue disorders) | 3 (3)
Superficial skin whitening after peel application (Skin and subcutaneous tissue disorders) | 6 (6)
Tingling (Skin and subcutaneous tissue disorders) | 6 (11)
Warm sensation (Skin and subcutaneous tissue disorders) | 4 (4)
Cold (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Earache (Ear and labyrinth disorders) | 1 (1)
Flu (Infections and infestations) | 1 (1)
Headache (General disorders) | 8 (8)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Menstrual pain (Endocrine disorders) | 4 (4)
Oedema (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore thorat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Stomachache (Gastrointestinal disorders) | 1 (1)
Toothache (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Increase in acne lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Inflammatory lump on right cheek after insect bite (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between Dermosciences France and the Clinical Research Organization who contracted the PI. Clinical Research Organization expressly agreed that any results communication must be submitted in advanced to Dermosciences France for approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT05821296/Prot_SAP_000.pdf